CLINICAL TRIAL: NCT03882034
Title: An Open-Label Phase 3 Study of the Safety and Efficacy of Pegvisomant in Children With Growth Hormone Excess
Brief Title: Safety and Efficacy of Pegvisomant in Children With Growth Hormone Excess
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190071; 19-CH-0071
Record Dates: First submitted 2019-03-19; First posted 2019-03-20 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11-04

CONDITIONS: Pituitary Disease
Keywords: Pediatric; Gigantism; Growth Hormone; Hormone; Pituitary Disease
MeSH Terms: conditions — Pituitary Diseases; Gigantism | interventions — pegvisomant

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Intervention arm, Patient received pegvisomant
  Interventions: Drug: Pegvisomant

INTERVENTIONS:
Drug: Pegvisomant — A fixed dose of pegvisomant 10-mg started on Day 1 of intervention and continued daily afterwards, will be administered subcutaneously according to manufacturer's recommendations. Adjustment of the dose will occur as per protocol.

SUMMARY:
Background:

For children with gigantism, too much growth hormone (GH) in the body causes abnormal growth and many other problems. Current treatments often don t work; no medical treatment is approved by FDA. Researchers want to see if the drug pegvisomant can help.

Objective:

To test the role of pegvisomant in children and adolescents with gigantism.

Eligibility:

People ages 2-18 with GH excess for whom usual treatments have not worked or who are not eliginle for them

Design:

Participants will be screened with a medical history.

The study will last 60 weeks and include at least 3 visits: baseline, 6-month, and 12-month visits. For the baseline visit, participants will stay a few nights for testing. They may stay overnight for the other visits.

All visits will include:

Medical history

Physical exam

Questionnaires

Heart and liver tests

Participants may be photographed in their underwear if they agree.

Blood tests: Participants will get a catheter: A small plastic tube will be placed in an arm vein. For some tests, the blood may be drawn every 30 minutes over 3 hours. For other tests, blood will be drawn every 20 minutes over 12 hours. Only clinically necessary tests will be done in each patient.

At the baseline visit, participants will have the study drug injected under the skin. They will learn to take the injection at home. They will take the injection daily during the study.

The baseline and 12-month visits will include:

MRI: Participants will have a dye injected into a vein. They will lie in a machine that takes pictures of the body.

Hand X-ray

Participants must get their height and weight at their local doctor s office monthly.

Participants must have blood and urine tests at their local lab monthly for the first 6 months then every 3 months until the study ends.

...

DETAILED DESCRIPTION:
Study Description:

GH excess is a rare and potentially lethal condition associated with hypersecretion of GH, usually by a pituitary tumor or hyperplasia. When it occurs prior to the complete fusion of growth plates, it leads to pathological tall stature, and it is called gigantism. After the fusion of the growth plates, it is called acromegaly. It may be associated with debilitating cardiovascular disease and/or diabetes. Children and adolescents with gigantism are currently treated with surgery, radiation therapy, and medications, such as octreotide, to reduce hypersecretion of GH; however, these treatments may lack efficacy and have significant side effects. Pegvisomant is a genetically engineered GH-receptor (GHR) antagonist that blocks the action of GH. In adults with acromegaly, pegvisomant has been shown to effectively reduce serum insulin-like growth factor type 1 (IGF-1) concentrations and lead to clinical improvement. However, experience in children and adolescents is limited to a small number of case series.,We propose the initiation of a new protocol at the NICHD, NIH, to treat children and adolescents with GH excess that is refractory to surgical therapy and/or radiation therapy, or in children and adolescents where the above therapies are contraindicated.

Objectives:

PRIMARY OUTCOMES:

* Percent change of IGF-1 z-score from baseline to end of study (12 month visit).
* Determine the safety and tolerability of pegvisomant in children and adolescents with GH excess.

SECONDARY OUTCOMES:

* Percent change of IGF-1 z-score from baseline to end of the study in subgroups of patients receiving monotherapy and patients receiving additional medication that target GH excess.
* Normalization of the IGF-1 for age and sex from baseline to end of study (normal value defined as +/- 2 SD from the mean). Change in growth velocity to a near-normal range (+/- 1 SD) according to the Tanner and Davies growth velocity curves for age, sex, and stage of puberty, when comparing the 6-month period prior to the study drug initiation to the growth velocity between 6 and 12 months on the study drug.
* Improvement in signs and symptoms of GH excess that are common in the pediatric population (headaches, excessive perspiration, fatigue, increased appetite) and the quality of life of the patients from baseline to the end of the study (12 month visit).
* Improvement of the cardiac structure and function: reduction of

the left ventricular mass index (LVMi), and change of the left

ventricular ejection fraction (EF) on echocardiogram from

baseline to the end of the study (12 month visit).

The objectives of the proposed study are to characterize the efficacy of pegvisomant as indicated by adequate control of the IGF-1 levels, the safety profile of the medication in children with GH excess, and to obtain pharmacodynamic data on the effect of pegvisomant on the GH-IGF axis in children. Because pegvisomant does not inhibit GH secretion, serum IGF-1 is the best marker of treatment efficacy. Pharmacokinetic (PK) studies will be performed in a subset of patients. This study will enroll patients with GH excess younger than 18 years and their biological parents.

Endpoints: Safety

Patients who have received at least 1 dose of pegvisomant will be included in the safety evaluations.

Safety will be evaluated by:

* Spontaneously reported adverse events
* Vital signs and periodic physical examinations (performed at the Clinical Center at baseline, 6 months (if possible unless telehealth visit performed) and 12 months after the study enrollment, and at local provider s office at regular intervals between those visits)
* Laboratory tests (performed periodically as indicated by previous studies) including:

  * Hematology
  * Chemistry
  * Lipids
  * Liver function panel
  * Thyroid function tests
  * IGF-1
  * Glucose and insulin
* MRI of the pituitary to check for tumor growth at baseline, 6 months, and 1 year
* Annual liver ultrasound
* ECG and echocardiogram at baseline, 6 months (EKG, if possible unless telehealth visit performed) and 1-year to monitor for the presence of cardiac arrhythmias and GH related cardiomyopathy
* Care providers will complete the Gigantism Symptoms Assessment Questionnaire (GSAQ) and Child Health Questionnaire by Landgraf & Wade for assessment of quality of life.
* Patients with gigantism and diabetes mellitus may require careful monitoring and dose reductions of insulin and/or oral hypoglycemic agents as pegvisomant usually has beneficial effects on glucose metabolism.7 Patients with pre-existing diabetes will continue to monitor their daily blood glucose levels, as previously instructed, and communicate with the investigational team for persistent elevation or decrease of the glucose levels. The changes of the dose of the anti-diabetic drugs and/or insulin will be done with communication of the research team with the local endocrinologist. Patients without pre-existing diabetes will be educated on the signs of hyperglycemia and will get monthly fasting blood glucose level measurements for the first 6 months along with the screening of the liver enzyme levels.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects who are eligible for enrollment must meet the following eligibility criteria:

Cohort 1: Patients with GH excess

* Males and females 24 months to <18 years at enrollment
* Active GH excess as demonstrated by the following:

  * IGF-1 greater than the upper limit of normal for age and sex during screening (>+2 SD) and
  * Abnormal GH levels as demonstrated by inability to suppress to <1 ng/mLwith older radioimmunoassays or <0.4ng/ml with sensitive immunoradiometric or immunochemiluminescent assays within 2 hours during Oral Glucose Tolerance Test (OGTT) after the administration of 1.75gr/kg (max 75gr) of glucose or elevated GH secretion profile during overnight sampling.
* History of inadequate response to trans-sphenoidal surgery or radiation therapy for GH secreting pituitary tumor, or inability to tolerate surgery or radiation therapies or patient deemed inappropriate candidate for surgery and/or pituitary radiation therapy, as determined by review of the medical records by the PI. The evaluation of the patient should be performed at 3 months after the surgery date in order to ensure that there is persistent GH excess after the transsphenoidal resection of the tumor unless there are clear evidence of persistent disease, e.g. residual tumor, based on the PI s assessment. If the patient has received irradiation, there is no minimum time to be considered before enrolling in the study. The effects of radiation therapy take place over many years after receiving it (mean time to remission for stereotactic radiation therapy of 12-60 months), and, thus, a medical therapy is required during that period.
* Patient is either not receiving any other medication for GH excess or is receiving stable dose/frequency of other medications for the treatment of GH excess prior to initiation of pegvisomant and no further adjustment or addition of new medication is made for the duration of the study.

  * Medications that may be co-administered for GH excess include but are not limited to: IM/SC/oral first- or second-generation somatostatin analogues (octreotide, lanreotide, pasireotide), oral dopamine agonist (cabergoline) and any other medication/formulation that may become available during this study. For each medication, its specific formulation and route of administration, patient will need to be on stable dose/frequency for a duration that is at least the minimum time recommended for adjusting the dose by the manufacturer which usually incorporates the time needed to reach plasma steady-state levels and a new plateau on the effect of the medication on IGF-1 (cabergoline: 4 weeks; SC octreotide/pasireotide administered twice or three times daily: 2 weeks; oral octreotide: 2 weeks; depot IM octreotide/SC lanreotide/IM pasireotide administered Q4 weeks: 3 months). The duration needed for the stable dose for patients on alternative schedules of administration of the above or other medications will be assessed based on available information and the longest estimated interval to achieve the full effect.
  * If a patient has been receiving a medication for GH excess but is not interested to continue that medication a minimum period of 6-weeks of discontinuation of the medication will be required for washout. This period was defined in the prior version of the protocol and is designed to minimize the time the patient may not be receiving any treatment for GH excess.
* Able to provide consent/assent if developmentally appropriate
* Willing to use non-hormonal method of contraception in patients of reproductive potential from the start of the study until at least 28 days after they stop the medication. Females of reproductive age (Tanner 3 or more, and/or having menstrual cycle) will be educated on the risks of unknown potential fetal harm while using the investigational medication, and they will be educated on the alternative preventative methods for contraception (condoms). Females already receiving oral contraceptive pills (OCPs) will be evaluated by gynecology consult service to discuss effective non-hormonal contraception. Sexually active female subjects must agree to use an effective non-hormonal contraception for the duration of the study.
* Have a primary health care provider in home location who will perform regular height and weight measurements, vital signs, and safety labs.

Height and weight will be requested to be performed according to the published methods included in the CDC-NHANES manual on anthropometry procedures manual (Supplementary Material). They will be plotted on the respective growth charts produced by the CDC for the US population (Supplementary Material).

Cohort 2: Parents

-Biological parents of a participant enrolled in the study enrolled for anthropometric measurements only.

EXCLUSION CRITERIA:

Cohort 1: Patients

An individual who meets any of the following criteria will be excluded from participation in this study:

* Liver function abnormalities (ALT, AST) greater than or equal to 3 x ULN
* Positive pregnancy test in females, current pregnancy and/or female patients who are breastfeeding.
* Patients currently using opioids. Opioids induce altered metabolism of pegvisomant. Since this is a phase 3 study, opioids may affect the PK studies to be performed and, thus, chronic use of opioids (>2 weeks) will be an exclusion criterion.
* Patients with any medical, physical, psychiatric, or social condition, which, in the opinion of the investigators, would make participation in this protocol not in their best interest, will be excluded from the study. Patients who are critically ill, unstable, or with severe organ failure that may affect/limit the endocrine evaluation and place unsustainable demands on CC or NICHD resources will be excluded.

Cohort 2: Patients Parents:

Subjects enrolled as parents of patients do not have to be tested for the above exclusion criteria as their participation is limited to anthropometric measurements (no risk).

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Percent change of IGF-1 z-score from baseline to end of study (12 month visit). | 1 year
  The primary endpoint is decrease in IGF-1 z-score >50% from baseline. This criterion will be used to determine efficacy.
Determine the safety and tolerability of pegvisomant in children with GH excess | During 1 year
  Safety will be determined by the periodical description of vital signs, laboratory and imaging studies, and other reported side effects.

SECONDARY OUTCOMES:
Normalization of IGF-1 for age and sex from baseline to end of study (12 month visit) | 1 year
  Normalization of the IGF-1 for age and sex from baseline to end of study (normal value defined as +/- 2 SD from the mean).
Normalization of growth velocity | 1 year
  Change in growth velocity to a near-normal range (+/- 1 SD) according to the Tanner and Davies growth velocity curves for age, sex, and stage of puberty, when comparing the 6-month period prior to the study drug initiation to the growth velocity between 6 and 12 months on the study drug.
Improvement in signs and symptoms of GH excess and quality of life from baseline to end of study (12 month visit) | 1 year
  Improvement in signs and symptoms of GH excess that are common in the pediatric population (headaches, excessive perspiration, fatigue, increased appetite) and the quality of life of the patients from baseline to the end of the study (12 month visit).
Left ventricular ejection fraction change on echocardiogram from baseline to end of study (12 month visit). | 1 year
  Improvement of the cardiac structure and function: reduction of the left ventricular mass index (LVMi), and change of the left ventricular ejection fraction (EF) on echocardiogram from baseline to the end of the study (12 month visit).
Reduction of the left ventricular mass index (LVMi) on echocardiogram from baseline to end of study (12 month visit) | 1 year
  (LVMi), and change of the left ventricular ejection fraction (EF) on echocardiogram from baseline to the end of the study (12 month visit).

CONTACTS AND LOCATIONS:
Overall Officials: Karim A Calis, Pharm.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Protocol is silent on IPD sharing.

REFERENCES:
- [Background] Trainer PJ, Drake WM, Katznelson L, Freda PU, Herman-Bonert V, van der Lely AJ, Dimaraki EV, Stewart PM, Friend KE, Vance ML, Besser GM, Scarlett JA, Thorner MO, Parkinson C, Klibanski A, Powell JS, Barkan AL, Sheppard MC, Malsonado M, Rose DR, Clemmons DR, Johannsson G, Bengtsson BA, Stavrou S, Kleinberg DL, Cook DM, Phillips LS, Bidlingmaier M, Strasburger CJ, Hackett S, Zib K, Bennett WF, Davis RJ. Treatment of acromegaly with the growth hormone-receptor antagonist pegvisomant. N Engl J Med. 2000 Apr 20;342(16):1171-7. doi: 10.1056/NEJM200004203421604. PMID 10770982
- [Background] Lodish MB, Trivellin G, Stratakis CA. Pituitary gigantism: update on molecular biology and management. Curr Opin Endocrinol Diabetes Obes. 2016 Feb;23(1):72-80. doi: 10.1097/MED.0000000000000212. PMID 26574647
- [Background] Katznelson L, Laws ER Jr, Melmed S, Molitch ME, Murad MH, Utz A, Wass JA; Endocrine Society. Acromegaly: an endocrine society clinical practice guideline. J Clin Endocrinol Metab. 2014 Nov;99(11):3933-51. doi: 10.1210/jc.2014-2700. Epub 2014 Oct 30. PMID 25356808
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-CH-0071.html